CLINICAL TRIAL: NCT02480127
Title: Molecular Evaluation of Endometrium Obtained From Women With Repeated Implantation Failure (RIF) After Endometrial Injury in Compare to Women Without Endometrial Injury; Phase 3 Clinical Trial
Brief Title: Molecular Evaluation of Endometrium After Endometrial Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: royan-Emb-021
Record Dates: First submitted 2015-06-07; First posted 2015-06-24 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Endometrial Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial injury (Experimental): In the intervention group, endometrial sampling is obtained twice by Pipelle [one in the follicular phase (during 8-9 or 11- 13 day in the beginning of buserelin cycle) and the last in the luteal phase (during 19-21 or 20-23 day) preceding the embryo transfer cycle preceding the embryo transfer cycle]. Blood samples (5- 10 cc) are taken in the both groups twice (one on the 9-8 or 11- 13 day and 19-21 or 20-23 day preceding the embryo transfer cycle).
  Interventions: Procedure: PIPELLE Endometrial injury
- Control (No Intervention): In the control group endometrial sampling will be done only in the luteal phase of the cycle preceding the embryo transfer cycle. Blood samples (5- 10 cc) are taken twice (one on the 9-8 or 11- 13 day and 19-21 or 20-23 day preceding the embryo transfer cycle).

INTERVENTIONS:
Procedure: PIPELLE Endometrial injury — The endometrial injury which is induced with pipelle.
  Arms: Endometrial injury

SUMMARY:
Repeated implantation failure (RIF) is determined when failure of implantation occurred during at least three consecutive IVF attempts while at least one high-grade embryo was transferred in each cycle. Several methods have been suggested to improve the implantation rate in RIF patients. One of the most promising methods is local injury to the endometrium. It has been reported that the rates of implantation, clinical pregnancy, and live birth reach more than double in RIF patients with local endometrial injury than patients without it. The population of this study included all infertile couples attending the Royan Institute, who have at least three consecutive cycles of ART failure. Also this study is phase 3 randomized clinical trial. Based on the average menstrual cycle 30-28 days, endometrial and blood samples were collected from two groups of patients on day 21 of luteal phase of their spontaneous menstrual cycle. The intervention, but not the control group underwent prior biopsy treatment in follicular phase on days 8 or/and 11 to 13 of that same cycle but in these days blood sample in both groups were collected. To investigate the impact of local endometrial injury in increasing the rate of pregnancy in ART - treated RIF patients, the investigators will examine the changes of immunological factors involved in the implantation including some cytokines, growth factors ( in serum and endometrial biopsies) and the expression of TLRs and HOX genes ( in endometrial biopsies) obtained from both groups.

DETAILED DESCRIPTION:
This study is phase 3 randomized clinical trial that the 20 infertile women with the following conditions will be studied in 2 groups. In the intervention group, Endometrial sampling is obtained twice by Pipelle [one in the follicular phase (during 8-9 or 11- 13 day in the beginning of buserelin cycle) and the last in the luteal phase (during 19-21 or 20-23 day) preceding the embryo transfer cycle preceding the embryo transfer cycle]. In the control group endometrial sampling will be done only in the luteal phase of the cycle preceding the embryo transfer cycle. Blood samples (5- 10 cc) are taken in the both groups twice (one on the 9-8 or 11- 13 day and 19-21 or 20-23 day preceding the embryo transfer cycle).

ELIGIBILITY:
Inclusion Criteria:

* < 40 years old
* Patients had history of 3 failed consecutive cycles of IVF / ICSI.
* Patients were good responders in prior ovulation induction cycle.
* There were at least two embryos with grade A in each embryo transfer cycle.
* Normal uterus in Hysterosalpingography (HSG) or ultrasound or hysteroscopy scans.
* The minimum thickness of the endometrium is 7 mm in injection day.

Exclusion Criteria:

* Submucosal myoma.
* Intramural and sub serousal myoma greater than 5 cm.
* Endometrioma equal to or greater than 3 cm or Hydrosalpinx.
* The number of available embryos is less than 2 in the current cycle.
* Patients with endometrial tuberculosis and persons who are treated for tuberculosis.
* Patients with any specific drug consumption.
* Patients with a history of thyroid disease, diabetes and other endocrine disorders.
* Lost to follow up or sampling.
* Impossibility of prepare endometrial sampling because of severe pain or probability infection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
cytokine | 1month
  Measurement of cytokines in endometrial sample in both group.
growth factor | 1month
  Measurement of growth factors in endometrial sample in both groups.

SECONDARY OUTCOMES:
Expression of TLRs | 1month
  Evaluation of TLRs expression in endometrial sample in both groups.
Expression of HOX | 1month
  Evaluation of HOX expression in endometrial sample in both groups.
pregnancy rate | 6months
  Evaluation of pregnancy rate in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Reza Aflatoonian, PhD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Centre, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Mahnaz Ashrafi, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Centre, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Samaneh Aghajanpour, M.S.c, Principal Investigator — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Centre, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Elham Amirchaghmaghi, MD,PhD, Principal Investigator — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Centre, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org